CLINICAL TRIAL: NCT06274671
Title: A Pilot Study to Investigate Glymphatic System Alterations in Vivo in Patients With Clinically Isolated Syndrome, Using Magnetic Resonance Imaging
Brief Title: Glymphatic MRI in Clinically Isolated Syndrome
Status: Recruiting | Type: Observational
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Other Study IDs: 23-24-09
Record Dates: First submitted 2024-01-31; First posted 2024-02-23 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Clinically Isolated Syndrome
Keywords: Clinically Isolated Syndrome; Multiple Sclerosis; Glymphatic System; Neuroimaging
MeSH Terms: conditions — Multiple Sclerosis | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples will be analyzed for biomarkers related to Clinically Isolated Syndrome and the function of the glymphatic system, and will be stored with consent for future analysis related to CIS/glymphatic system research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Clinically Isolated Syndrome: Patients with a diagnosis of Clinically Isolated Syndrome
  Interventions: Other: Magnetic Resonance Imaging
- Healthy Controls: Age- and gender-matched healthy controls.
  Interventions: Other: Magnetic Resonance Imaging

INTERVENTIONS:
Other: Magnetic Resonance Imaging — A Magnetic Resonance Imaging (duration: about 60 minutes) with research sequences for the visualization of alterations of the glymphatic system.

SUMMARY:
The brain possesses a system to get rid of unwanted substances, named Glymphatic System (GS). When this system is faulty, these accumulate, there is local inflammation, and progressive death of the cells. This occurs in neurological diseases including Parkinson's, or Alzheimer's. Inflammation and progressive death of the cells are also present in another neurological disorder, named Multiple Sclerosis (MS).

Doctors think that GS dysfunction plays a role in MS too. In this research therefore, the aim is to study whether it drives inflammation, and disease progression in MS patients.

The researchers have developed a new way to find signs of alteration of the GS using a scan named Magnetic Resonance Imaging (MRI) and will use it in a pilot study on patients with a condition named Clinically Isolated Syndrome (CIS), which often represents the very beginning of MS. It would therefore be demonstrated that the GS is a new mechanism of disease in CIS, which may associate with the symptoms, or the alterations in the levels of some substances in the blood suggestive of brain cells damage.

Should this study be successful, this would provide preliminary evidence to perform a larger research study to assess if GS dysfunction drives the progression of MS.

DETAILED DESCRIPTION:
This is a cross-sectional case-control study on patients with a diagnosis of Clinically Isolated Syndrome (CIS) and a group of age- and gender-matched healthy controls.

In this study all participants will undergo two visits. In the first visit, all participants will sign the informed consent form and perform a detailed neurological examination, with administration of a few questionnaires for assessment of symptoms related to CIS/Multiple Sclerosis. Participants will also donate a sample of blood for safety analysis, analysis of biomarkers related to CIS and the glymphatic system, as well as for storage in a biobank. Participants will donate a sample of urine for urinalysis and pregnancy test in females of childbearing potential.

In the second visit, all participants will visit the Mireille Gillings Neuroimaging Centre of the University of Exeter for an MRI scan, that will last about 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 or over
2. Suitable physically and psychologically to undertake the assessments, as judged by the Investigator
3. Have voluntarily provided informed consent and have signed an ICF indicating that the purpose of the study has been explained and are willing and able to adhere to the study procedures described in the ICF.
4. (For CIS group): A diagnosis of CIS or MS at first presentation
5. Subjects must not have taken corticosteroids or IVIg or plasma-exchange within the 30 days prior to consent
6. Adequate vision and hearing to perform the study procedures
7. Medically healthy with no clinically significant findings on physical examination, laboratory profiles, vital signs at screening (with the exception of the signs of the condition under investigation)
8. Women of child-bearing potential must practice a medically acceptable method of birth control. Acceptable methods include oral contraceptive, contraceptive patch, long-acting injectable contraceptive, or double-barrier method (condom or intrauterine device with spermicide).
9. If on immunomodulatory medication, patients must have started it at least 30 days from screening and should not change their medication dose for the duration of the study.

Exclusion Criteria:

1. Have a diagnosis of clinically definite Multiple Sclerosis according to the 2017 McDonald's Criteria (Thompson et al., 2018)
2. Have a CIS limited to the spinal cord (transverse myelitis)
3. Present psychiatric disorders or severe cognitive deficit
4. Past or present history of drug or alcohol abuse
5. Are pregnant or breastfeeding, if females of childbearing potential
6. Have any other medical, neurological, or psychiatric condition or clinically significant laboratory abnormality excluding CIS which, in the opinion of the Investigator, might preclude participation
7. Are taking benzodiazepines on a regular basis or are unable to suspend intake of benzodiazepines
8. Have received any investigational product within a time-period equal to five half-lives of the product, if known, or minimum of 60 days before consent
9. Are unable to lie down for MRI scanning
10. Have any finding on the brain MRI that would compromise subject safety or the scientific integrity of the study
11. Have implants, such as implanted cardiac pacemakers or defibrillators, insulin pumps, cochlear implants, metallic ocular foreign body, implanted neural stimulators, aneurysm clips, or other medical implants that have not been deemed safe for MRI
12. Have a history of claustrophobia
13. Have any other contraindication to MRI scanning
14. Have a relapse occurred after consent but before the MRI scan
15. It is preferable the following laboratory tests are part of the subject's medical history for differential diagnosis of clinically isolated syndrome (CIS): erythrocyte sedimentation rate (ESR), antinuclear antibody (ANA), complement (C3, C4) and anticardiolipin IgG - IgM

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1: Patients with a diagnosis of Clinically Isolated Syndrome Group 2: Healthy controls
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine that patients with CIS display alterations of the glymphatic system visible in vivo by Structural MRI | Through study completion, an average of 7 days
  Difference between CIS and HV in the number of perivascular spaces
To determine that patients with CIS display alterations of the glymphatic system visible in vivo by microstructural MRI | Through study completion, an average of 7 days
  Difference between CIS and HV in estimation of intraparenchymal water transport
To determine that patients with CIS display alterations of the glymphatic system visible in vivo by diffusion-weighted MRI | Through study completion, an average of 7 days
  Difference between CIS and HV in the calculation of the ALPS-index
To determine that patients with CIS display alterations of the glymphatic system visible in vivo by perfusion-MRI | Through study completion, an average of 7 days
  Difference between CIS and HV in estimation of choroid plexus perfusion
To determine that patients with CIS display alterations of the glymphatic system visible in vivo by ALS-MRI | Through study completion, an average of 7 days
  Difference between CIS and HV in estimation of Cerebrospinal Fluid (CSF) flow

SECONDARY OUTCOMES:
To correlate in vivo measures of altered glymphatic system with MRI measures of structural integrity in CIS | Through study completion, an average of 7 days
  Quantification in CIS of structural volumetric and thickness
To correlate in vivo measures of altered glymphatic system with MRI measures of disease activity in CIS | Through study completion, an average of 7 days
  Quantification in CIS of total lesion load
To correlate in vivo measures of altered glymphatic system with MRI measures of enlarged Wirchow-Robin spaces in CIS | Through study completion, an average of 7 days
  Quantification in CIS of perivascular spaces
To correlate in vivo measures of altered glymphatic system with MRI measures of microstructural altertions in CIS | Through study completion, an average of 7 days
  Quantification in CIS of free water, a measure of extracellular space
To correlate in vivo measures of altered glymphatic system with MRI measures of brain perfusion in CIS | Through study completion, an average of 7 days
  Quantification in CIS of water transport and regional perfusion.
To correlate in vivo measures of altered glymphatic system in CIS with clinical measures of disease severity | Through study completion, an average of 7 days
  Correlation between MRI measures and EDSS score in CIS patients.
To correlate in vivo measures of altered glymphatic system in CIS with fluid biomarkers of axonal injury in CIS | Through study completion, an average of 7 days
  Correlation between MRI measures and fluid biomarkers for neuroaxonal integrity (calculated with the quantification of Neurofilament Light Chain (NfL)
To correlate in vivo measures of altered glymphatic system in CIS with fluid biomarkers of astrocytis integrity in CIS | Through study completion, an average of 7 days
  Correlation between MRI measures and fluid biomarkers for astrocytic activation (calculated with the quantification of Glial Fibrillary Acid Protein (GFAP)
To correlate in vivo measures of altered glymphatic system in CIS with fluid biomarkers of glymphatic activity in CIS | Through study completion, an average of 7 days
  Correlation between MRI measures and fluid biomarkers for glymphatic transport damage (calculated with the quantification of Aquaporin 4 (AQP4) and of Neuronal-Specific Enolase (NSE)

CONTACTS AND LOCATIONS:
Overall Officials: Edoardo R de Natale, MD, Principal Investigator — University of Exeter
Locations (2):
- United Kingdom (2):
  - University of Exeter, Exeter, Exeter
  - Royal Devon University Healthcare NHS Foundation Trust, Exeter

IPD SHARING:
Plan to Share IPD: No